CLINICAL TRIAL: NCT07352033
Title: Is Pulse Co-Oximetry a Reliable Alternative to Invasive Hemoglobin Measurement in Pediatric Neurosurgical Procedures?
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, FUNDA ARUN, Assistant Professor, Selcuk University
Other Study IDs: F6
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anemia (Diagnosis)
MeSH Terms: conditions — Anemia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pediatric Neurosurgery Patients: Pediatric patients undergoing neurosurgical procedures requiring invasive arterial pressure monitoring and hemoglobin measurement
  Interventions: Device: Masimo Radical-7® Pulse CO-Oximeter

INTERVENTIONS:
Device: Masimo Radical-7® Pulse CO-Oximeter — Continuous non-invasive measurement of total hemoglobin (SpHb) using a pulse co-oximetry sensor during the surgery.

SUMMARY:
The study evaluated the diagnostic accuracy and clinical utility of continuous SpHb across a comprehensive pediatric age spectrum-ranging from neonates to adolescents-undergoing high-risk neurosurgical procedures (cranial and spinal) characterized by significant potential for blood loss.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-IV,
* Scheduled for elective complex spinal surgery or cranial procedures under general anesthesia

Exclusion Criteria:

* congenital heart disease
* requirement for emergency surgery
* pre-existing peripheral circulatory disorders

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients admitted to the Department of Neurosurgery for elective surgery requiring general anesthesia and invasive arterial blood pressure monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Agreement and Correlation between Non-invasive Hemoglobin (SpHb) and Invasive Arterial Hemoglobin (Hb) levels. | Intraoperative period (from induction of anesthesia to extubation, approximately 2-5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided